CLINICAL TRIAL: NCT06166940
Title: Comparison Of The Two Types Of Hemostasis Management Effectiveness : Thromboelastometry (Rotem) Guided Management And Conventional Method In Newborn Congenital Cardiac Surgery Patients
Acronym: hemostasis
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023.11.11
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-03

CONDITIONS: Newborn Cardiac Surgery; Newborn Hemostasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conventional Management
  Interventions: Other: ROTEM Guided Management

INTERVENTIONS:
Other: ROTEM Guided Management — ROTEM guided management of hemostasis after CPB

SUMMARY:
Sixty consecutive newborn patients who underwent pediatric cardiac surgery from April 2022 to October 2023 at Basaksehir Cam and Sakura City Hospital) were included in this study. Data of eighty-six patients who received ROTEM guided transfusions after August 15, 2022 was collected. First sixteen patients were given cryoprecipitate in the middle of the Modified ultra-filtration (MUF) procedure according to previous conventional approach, and so these patients excluded. And ten patients were excluded due to the lack of information. Thirty patients, who received ROTEM guided transfusions compared to the prior thirty patients who received transfusions conventionally. There was no randomization and standardized anesthesia and surgical techniques were used.

Anesthesia induction conducted with midazolam, ketamine, fentanyl, and rocuronium bromide; and antifibrinolytic (tranexamic acid) infusion was used during operation till the closure of skin. Anesthesia and cardiopulmonary bypass(CPB) anesthesia was maintained with remifentanil, midazolam, ketamine and rocuronium, and sevoflurane -not during bypass. Size-adapted bypass circuits and membrane oxygenators (FX05 oxygenators) were used. Total priming volume for the bypass circuit was 250 - 400 ml, consisting of red blood cell (RBC), fresh frozen plasma (FFP), Isolyte-S solution, mannitol, sodium bicarbonate, tranexamic acid, prednisol, and antibiotic. Anticoagulation during CPB was managed with 350 U/kg unfractioned heparin (Novo-Heparin) and additional boluses of 50 U/kg, as needed, to maintain an activated clotting time (ACT) of at least 450s. Heparin anticoagulation was antagonized with 3,5 mg/kg protamine.

Red blood cell concentrates were transfused to maintain the haematocrit at 28 - 32% during cardiopulmonary bypass (CPB). Bypass was conducted under mild (core temperature 32°C ) and moderate (core temperature 28 °C) hypothermia. Myocardial protection was achieved with cold intermittent blood cardioplegia (20 ml/kg), which was prepared during CPB by adding buffered del nido solution (Plasma-Lyte A) in the ratio 1:4 to whole blood obtained from the arterial line. The cardioplegia solution was kept at 6°C before infusion. Blood sample for running ROTEM analysis were taken just before weaning CPB, when the core temperature of patients were 36-37 °C. MUF was performed after weaning from CPB and 5-10 minutes before protamine administration, with a target haematocrit of 35-40%. After heparin antagonization, RBC transfusions applied with a target haematocrit of 35-40 % for non-cyanotic patients, and 40-45% for cyanotic patients.

We collected data on the following subject characteristics: height (cm); weight (kg); age (days); gender; presence of cyanosis; presence of ay genetic disorder; Aristotle score (1,5-25); duration of the surgical procedure (min); CPB time (min); aortic cross clamp time (min); the lowest core temperature during CPB; total amount of blood products transfused after CPB intraoperatively (ml/kg), including red blood cell concentrates, FFP, platelet concentrates, cryoprecipitate, and fibrinogen concentrates; total amount of blood products transfused after operation up to 24 h after admission to the Pediatric Cardiac Intensive Care Unit (PCICU) (ml/kg); total amount of chest tube drainage after operation up to 24 h after PCICU admission (ml/kg); 28 day survival; extracorporeal membrane oxygenator (ECMO) application; and need for peritoneal dialysis.

In all patients, routine blood samples for hemoglobin (Hb), haematocrit (Hct), prothrombin time (PT), international normalized ratio (INR), activated partial thromboplastin time (aPTT), platelet count; renal function tests urea and creatinine were collected preoperatively. Hb, Hct, PT, INR, aPTT, platelet count, urea and creatinine were also analyzed on the first postoperative morning.

We conducted thromboelastometry in the operating theatre (OR) using the ROTEM device. Four assays-EXTEM, INTEM, FIBTEM, and HEPTEM were tested in citrated whole blood. Because the patients were still under heparin effect when the samples were taken, we made transfusion adjustments according to EXTEM and FIBTEM test results. Since we got the EXTEM, FIBTEM A5 results as soon as heparin antagonization was complete, we transfused the blood products according to the results. We also collected those data.

The primary outcome was the proportion of perioperative transfusion (intraoperatively and in the PCICU) in the ROTEM group and in the conventional group. The secondary outcomes are postoperative chest tube drainage up to 24 hours; need for peritoneal dialysis. The other analyses have mainly a descriptive purpose.

DETAILED DESCRIPTION:
Four main scenarios based on clinical observation and ROTEM results were possible:

1. Insignificant bleeding-normal ROTEM; no transfusions
2. Insignificant bleeding-abnormal ROTEM; no transfusions
3. Significant bleeding-normal ROTEM; surgical reevaluation
4. Significant bleeding-abnormal ROTEM; transfusion of blood products as indicated by:

   1. FIBTEM A5 <9 mm -fibrinogen concentrate or cryoprecipitate
   2. 9mm ≤ FIBTEM A5 <13mm and or EXTEM CT > 80 seconds fibrinogen concentrate or cryoprecipitate and significant bleeding still continued with EXTEM A5 < 35 mm - platelet concentrate
   3. FIBTEM A5 >13mm and EXTEM A5 < 35 mm -platelet concentrate
   4. After transfusions if the bleeding was still continuing, while surgical reevaluation was in progress, we gave fibrinogen concentrate to replace the lost fibrinogen with the ongoing bleeding. At the same time to verify the treatment effect and control heparin reversal, a second set of INTEM, HEPTEM, EXTEM and FIBTEM analyses were also performed during wound closure. ACT was tested in all patients to control for heparin reversal. If patients had both a pathological ACT and ROTEM (CTIN/ CTHEP ratio ≥ 1,25) protamine was administered first. After fibrinogen and platelet transfusions, if INTEM CT > 280 seconds and HEPTEM CT > 280 seconds with continuing bleeding FFP were given.

Blood transfusion after paediatric intensive care unit (PCICU) admission was managed without ROTEM guidance by paediatric cardiac surgeons and intensivists.

ELIGIBILITY:
Inclusion Criteria:

* newborn patients who underwent pediatric congenital heart surgery on cardiopulmonary bypass

Exclusion Criteria:

* the newborn patients who did not need cardiopulmonary bypass during surgery were excluded.
* the newborns whose records are missing were excluded

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn patients who underwent pediatric congenital heart surgery on cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
perioperative transfusion | after weaning from cardiopulmonary bypass up to the end 24 hours
  the proportion of perioperative transfusion of RBC, fibrinogen concentrate, platelet concentrate, FFP in milliliters

SECONDARY OUTCOMES:
postoperative bleeding | from the admission of the pediatric cardiac intensive care unit up to 24 hours
  postoperative chest tube drainage in milliliters

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)